CLINICAL TRIAL: NCT03864861
Title: Postoperative Outcomes Within an Enhanced Recovery After Bariatric Surgery Protocol POWER3
Brief Title: Postoperative Outcomes Within an Enhanced Recovery After Bariatric Surgery Protocol
Acronym: POWER3
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Grupo Español de Rehabilitación Multimodal (Other)
Collaborators: Sociedad Española de Cirugía de la Obesidad (Unknown); REDGERM (Unknown)
Responsible Party: Sponsor
Other Study IDs: REDGERM04
Record Dates: First submitted 2019-03-04; First posted 2019-03-06 (Actual); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: Perioperative Care; Postoperative Complications; Bariatric Surgery Candidate
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Elective Bariatric Surgery: Patients older than 18 undergoing elective bariatric surgery

SUMMARY:
Methods National audit of a 90-day prospective observational cohort in which pre-defined postoperative complications were analyzed at 30 days of follow-up in adult patients undergoing elective bariatric surgery with or without an intensified recovery program (ERAS: Enhanced Recovery after Surgery) with any level of protocol compliance (0-100%)

Research Places Spanish Hospitals where this surgical intervention is carried out.

Objectives To determine the incidence of postoperative complications per patient and procedure, regardless of the degree of adherence to ERAS protocols and its impact on the hospital stay and postoperative complications including 30-day mortality.

Sample size For an alpha error of 5% (95% confidence) and an accuracy of 3% and estimating a number of patients with complications of 11%, the sample size calculation yields 460 patients, although the final sample size it may be smaller depending on the proportion of complications detected.

Inclusion criteria Patients older than 18 years who are going to be electively operated on for bariatric surgery regardless of their adherence to an ERAS intensified recovery program and the compliance level of the protocol (from 0-100%)

Statistical analysis Continuous variables will be described as mean and standard deviation, if it is a normal distribution, or median and interquartile range, if they are not normally distributed. Comparisons of continuous variables will be performed by one-way ANOVA or the Mann-Whitney test, as appropriate. A univariate analysis will be performed to test the factors associated with postoperative complications, hospital stay and death in the hospital. Univariate analyzes and hierarchical multivariate logistic regression models will be constructed to identify factors associated independently with these results and to adjust for differences in confounding factors. The factors will be introduced in the models based on their relationship with the univariate result (p <0.05), the biological plausibility and the low rate of missing data.

DETAILED DESCRIPTION:
The results of this study will allow to identify, on the one hand, the type of patients presenting postoperative complications and, on the other hand, to identify those items of the ERAS protocols that are independently associated with a reduction in postoperative complications and hospital stay, which will allow to focus the perioperative efforts in those items that actually improve the postoperative outcomes.

Aim 1 will establish the number of patients developing predefined postoperative complications within 30 days of surgery in adult patients undergoing elective bariatric surgery with any compliance of an ERAS protocol (including patients with 0 compliance). This will allow us to determine the actual impact of these protocols.

Aim 2 will allow us to know the type of predefined complication presented by the patients included in the ERAS protocols and in patients undergoing bariatric surgery; This will allow, on the one hand, to have a starting point for future clinical trials, and, on the other hand, to focus efforts to avoid these complications.

Aim 3 will allow us to identify those perioperative items of ERAS protocols that are actually associated with a decrease in postoperative complications.

The proposed study will establish a real view of the number of patients presenting postoperative complications that will overcome the limitations of available retrospective studies and provide greater insight into the items of the protocols that are associated with decreased complications; on the other hand, the investigator's hypothesis is that the number of patients who develop predefined postoperative complications within 30 days of surgery decreases as there is greater compliance with the predefined ERAS protocol items

ELIGIBILITY:
Inclusion Criteria:

* All adult patients (aged ≥18 years) undergoing elective bariatric surgery and by any approach (Includes surgery with laparoscopic, assisted laparoscopic approach or open approach) in a participating hospital during the 30-day cohort period with a planned overnight stay.

Exclusion Criteria:

* Patients undergoing emergency surgery

  * Endoscopic procedures
  * Patients under 18 years of age
  * Patients with previous bariatric surgery who undergo revision surgery
  * Patients who refuse to participate

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients (aged ≥18 years) undergoing elective bariatric surgery
Sampling Method: Non-Probability Sample
Enrollment: 460 (Estimated)
Dates: Start 2019-10-22 (Estimated); Primary Completion 2020-02-22 (Estimated); Study Completion 2020-03-22 (Estimated)

PRIMARY OUTCOMES:
Predefined mild-moderate-severe postoperative complications | 30 days after surgery
  Standards for definitions and use of outcome measures for clinical effectiveness research in perioperative medicine were published by the European Perioperative Clinical Outcome (EPCO) definitions. Infectious complications, cardiovascular complications and other types of complications. Each complication will be graded as mild, moderate or severe.

SECONDARY OUTCOMES:
In-hospital all-cause mortality | 30 days after surgery
  The percentage of deaths within 30 days of surgery will be reported for each surgical category
ERAS Compliance | 30 days after surgery
  Overall compliance will be calculated as the average of all pre- and intraoperative ERAS adapted elements, as specified in the ERAS society bariatric guidelines ERAS patients' guideline compliance will be categorised into quartiles
Duration of hospital stay | 30 days after surgery
  The median hospital length of stay (LOS) following the start of surgery, overall, by survival status and by complication status will be reported. Post-operative LOS is the duration in days from the date of the end of surgery to the date of discharge from hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Javier M Ripollés-Melchor, Study Chair — Infanta Leonor University Hospital, Madrid, Spain; Raquel M Sanchez Santos, Study Chair — Complejo Hospitalario Universitario de Vigo; José M Ramírez, Study Director — Lozano Blesa University Hospital, Zaragoza, Spain; Jaime Ruiz Tovar, Study Director — Hospital Universitario Rey Juan Carlos Móstoles, Spain; César Aldecoa, Study Director — Hospital Universitario Río Hortega, Valladolid, Spain; Carlos Ferrando-Ortolá, Study Director — Hospital Clinic of Barcelona; Ester Martín García-Almenta, Study Director — Hospital Universitario Clínico San Carlos, Madrid; Ane Abad-Motos, Study Director — Infanta Leonor University Hospital, Madrid, Spain; Alfredo Abad-Gurumeta, Study Director — Infanta Leonor University Hospital, Madrid, Spain; Alejandro Suárez de la Rica, Study Director — Hospital Universitario La Paz
Locations (53):
- Spain (53):
  - Hospital Virgen de los Lirios de Alcoy, Alcoy, Alicante
  - Hospital General Universitario de Elche, Elche, Alicante
  - Hospital de Mérida, Mérida, Badajoz
  - Hospital Universitario Parc Tauli, Sabadell, Barcelona
  - Hospital de Sant Joan Despí Moisès Broggi, Sant Joan d'Espi, Barcelona
  - Hospital Universitario de Vic, Vic, Barcelona
  - Hospital Universitario de Cruces, Barakaldo, Bizkaia
  - Hospital General Universitario de Castellón, Castellon, Castellón
  - Complejo Hospitalario Universitario de A Coruña, A Coruña, Coruña
  - Hospital Universitario Puerta del Mar, Cadiz, Cádiz
  - Hospital Universitario Jerez de La Frontera, Jerez de la Frontera, Cádiz
  - Hospital Universitario Príncipe de Asturias, Alcalá de Henares, Madrid
  - Hospital Universitario Fundación Alcorcón, Alcorcón, Madrid
  - Hospital Universitario de Fuenlabrada, Fuenlabrada, Madrid
  - Hospital Universitario Getafe, Getafe, Madrid
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid
  - Hospital Rey Juan Carlos, Móstoles, Madrid
  - Hospital Universitario de Móstoles, Móstoles, Madrid
  - Hospital Universitario Quirón Madrid, Pozuelo de Alarcón, Madrid
  - Hospital Universitario de Torrejón, Torrejón de Ardoz, Madrid
  - Hospital General Mateu Orfila, Menorca, Menorca
  - Hospital Costa del Sol, Marbella, Málaga
  - Hospital Universitario Virgen del Victoria de Málaga, Málaga, Málaga
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Clínic Universitat de Barcelona, Barcelona
  - Hospital Universitario Sant Pau, Barcelona
  - Hospital Universitario Vall d´Hebrón, Barcelona
  - Hospital Universitario de Burgos, Burgos
  - Hospital General Universitario de Ciudad Real, Ciudad Real
  - Hospital Universitario de Guadalajara, Guadalajara
  - Hospital Universitario de Gran Canaria Doctor Negrín, Las Palmas
  - Hospital Universitario Insular de Gran Canaria, Las Palmas de Gran Canaria
  - Hospital Clínico San Carlos, Madrid
  - Hospital de La Princesa, Madrid
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Infanta Leonor, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital General Universitario José María Morales Messeguer, Murcia
  - Complejo Hospitalario y Universitario de Pontevedra, Pontevedra
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Universitario Virgen de Valme, Seville
  - Hospital Universitario Virgen Macarena, Seville
  - Complejo Hospitalario de Toledo, Toledo
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital General Universitario de Valencia, Valencia
  - Hospital Universitario La Fe, Valencia
  - Hospital Clínico de Valladolid, Valladolid
  - Hospital Universitario Río Hortega, Valladolid
  - Hospital Universitario de Álava, Vitoria-Gasteiz
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza
  - Hospital Universitario Miguel Server, Zaragoza

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ripolles-Melchor J, Sanchez-Santos R, Abad-Motos A, Gimeno-Moro AM, Diez-Remesal Y, Jove-Albores P, Arago-Chofre P, Ortiz-Sebastian S, Sanchez-Martin R, Ramirez-Rodriguez JM, Trullenque-Juan R, Valenti-Azcarate V, Ramiro-Ruiz A, Correa-Chacon OC, Batalla A, Gimeno-Grauwinkel C, Sanahuja-Blasco JM, Gonzalez-Valverde FM, Galan-Menendez P, Diez-Zapirain MJ, Vilallonga R, Zorrilla-Vaca A, Pascual-Bellosta AM, Martinez-Ubieto J, Carrascosa-Miron T, Ruiz-Escobar A, Martin-Garcia-Almenta E, Suarez-de-la-Rica A, Bausili M, Palacios-Cordoba A, Olvera-Garcia MM, Meza-Vega JA, Sanchez-Pernaute A, Abad-Gurumeta A, Ferrando-Ortola C, Martin-Vaquerizo B, Torres-Alfonso JR, Aguado-Sanchez S, Sanchez-Cabezudo-Noguera F, Garcia-Erce JA, Aldecoa C; POWER 3 Study Investigators Group. Higher Adherence to ERAS Society(R) Recommendations is Associated with Shorter Hospital Stay Without an Increase in Postoperative Complications or Readmissions in Bariatric Surgery: the Association Between Use of Enhanced Recovery After Surgery Protocols and Postoperative Complications after Bariatric Surgery (POWER 3) Multicenter Observational Study. Obes Surg. 2022 Apr;32(4):1289-1299. doi: 10.1007/s11695-022-05949-6. Epub 2022 Feb 10. PMID 35143011